CLINICAL TRIAL: NCT07035977
Title: A Deep-learning System for Low-Dose CBCT Image Reconstruction: a Stepwise, Multicentre, Early-stage Clinical Validation Study
Brief Title: DeepPriorCBCT for Low Dose Lung CBCT Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: DeepPriorCBCT001
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Lung Nodules
Keywords: DeepPriorCBCT; Lung nodules; Low dose radiation; Cross-Over Observational Study; CBCT; Percutaneous thoracic biopsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants will receive a 1/6 views undersampling lung CBCT scan. (Experimental): Participants will receive a 1/6 views undersampling lung CBCT scan. And the CBCT images will be reconstructed by DeepPriorCBCT model for further analysis.
  Interventions: Radiation: Participants will receive a 1/6 views undersampling lung CBCT scan.
- Participants will receive a full-sampling lung CBCT scan. (No Intervention): Participants will receive a full-sampling lung CBCT scan. And the CBCT images will be reconstructed by current clinical method for further analysis.

INTERVENTIONS:
Radiation: Participants will receive a 1/6 views undersampling lung CBCT scan. — Participants will receive a 1/6 views undersampling lung CBCT scan. And the CBCT images will be reconstructed by DeepPriorCBCT model for further analysis.
  Arms: Participants will receive a 1/6 views undersampling lung CBCT scan.

SUMMARY:
The goal of this clinical trial is to learn if the DeepPriorCBCT model ensure high-quality CBCT image while reducing CBCT radiation dose. The main questions it aims to answer are:

* Can DeepPriorCBCT reduce CBCT radiation doses?
* Is the image quality of DeepPriorCBCT reconstruction consistent with that of existing clinical reconstruction method? Researchers will compare CBCT images quality reconstruction with DeepPriorCBCT model to CBCT image quality reconstruction with existing clinical protocols to see if DeepPriorCBCT model can improve the CBCT image quality while reducing radiation dose.

Participants will:

* Receive a single low dose (1/6 of existing clinical protocols) CBCT scan
* Receive a single conventional dose CBCT scan

ELIGIBILITY:
Inclusion Criteria:

1. Participants will receive percutaneous thoracic puncture under the guidance of CBCT during the study period.
2. The participants' medical records containing basic information, medical history, etc are complete.
3. Participants can understand the study's purpose, procedures, potential risks, and benefits, and voluntarily signs a written informed consent form.

Exclusion Criteria:

1. Participants are under the age of 18.
2. Participants are suffering from severe mental illness or cognitive impairment, unable to understand the study and sign.
3. Participants are pregnant or breastfeeding women.
4. Participants are concurrent participating in other programs that affect the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
CBCT Images Quality Score | No more than 1 week
  CBCT Images Quality Score was analyzed by 5 radiologists using 5-point Likert scale.

SECONDARY OUTCOMES:
The scores of lesion diagnosis from 5 radiologists | No more than 1 week
  5 radiologists from 5 medical centers will be invited to diagnosis the lesion of fully sampled machine-reconstructed CBCT images vs. undersampled model-reconstructed CBCT images.
The agreement scores given by the 25 interventionalists. | No more than 1 week.
  25 interventionalists from 5 medical centers will be invited to analyze fully sampled machine-reconstructed CBCT images vs. undersampled model-reconstructed CBCT images. The scores given by the 25 interventionalists will be used for agreement score analysis.
Radiation dose | No more than 1 day
  Radiation dose is defined as the radiation dose received by patients when undergoing one conventional-dose CBCT scan and one undersampled CBCT scan.

OTHER OUTCOMES:
Objective indicators for reconstructed CBCT images | No more than 1 week.
  Objective indicators for reconstructed CBCT images include peak signal to noise ratio (PSNR) and structure similarity (SSIM). PSNR is a ratio that represents the ratio between the maximum possible power of a signal and the destructive noise power that affects its representation accuracy. SSIM is a metric for measuring image similarity.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The First Affiliated Hospital East Campus of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Wuhan Union Jinyin Lake Hospital, Wuhan, Hubei
  - Wuhan Union West Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bosch de Basea M, Thierry-Chef I, Harbron R, Hauptmann M, Byrnes G, Bernier MO, Le Cornet L, Dabin J, Ferro G, Istad TS, Jahnen A, Lee C, Maccia C, Malchair F, Olerud H, Simon SL, Figuerola J, Peiro A, Engels H, Johansen C, Blettner M, Kaijser M, Kjaerheim K, Berrington de Gonzalez A, Journy N, Meulepas JM, Moissonnier M, Nordenskjold A, Pokora R, Ronckers C, Schuz J, Kesminiene A, Cardis E. Risk of hematological malignancies from CT radiation exposure in children, adolescents and young adults. Nat Med. 2023 Dec;29(12):3111-3119. doi: 10.1038/s41591-023-02620-0. Epub 2023 Nov 9. PMID 37946058
- [Result] Mazzone PJ, Lam L. Evaluating the Patient With a Pulmonary Nodule: A Review. JAMA. 2022 Jan 18;327(3):264-273. doi: 10.1001/jama.2021.24287. PMID 35040882